CLINICAL TRIAL: NCT05960591
Title: Usability of the ADEPTH Sensor for Bore Depth Measurements in Plate Osteosynthesis Procedures: a Monocenter Randomized Pilot Study
Brief Title: Usability of the ADEPTH Sensor for Bore Depth Measurements in Plate Osteosynthesis Procedures
Acronym: ADEPTH-Pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SLAM Ortho B.V. (Industry)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MEC-2023-0269
Record Dates: First submitted 2023-07-07; First posted 2023-07-27 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Fractures, Bone; Osteosynthesis
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in either the control group (bore depth measurement with the manual depth gauge) or in the intervention group (bore depth measurements with the ADEPTH sensor).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants will receive bore depth measurements with the manual depth gauge, which is the golden standard for bore depth measurements during plate osteosynthesis procedures.
- Intervention (Experimental): Participants will receive bore depth measurements with the ADEPTH sensor, which is a new sensor technology for bore depth measurements during plate osteosynthesis procedures.
  Interventions: Device: ADEPTH

INTERVENTIONS:
Device: ADEPTH — ADEPTH sensor will be used for bore depth measurements during plate osteosynthesis procedures.
  Other Names: ADEPTH sensor
  Arms: Intervention

SUMMARY:
The goal of this monocenter randomized pilot study is to investigate the usability of the ADEPTH sensor for bore depth measurements in plate osteosynthesis procedures. The main question it aims to answer is:

- What is the usability score of the ADEPTH sensor for bore depth measurements during plate osteosynthesis procedures? Participants will receive either bore depth measurements with the ADEPTH sensor or with the manual depth gauge.

DETAILED DESCRIPTION:
To assess the usability score of the ADEPTH sensor for bore depth measurements in plate osteosynthesis procedures. The surgeon and OR-assistant will fill in one survey after performing 3 operations with the ADEPTH sensor and one survey after performing 3 operations with the manual depth gauge.

ELIGIBILITY:
Inclusion Criteria:

* Elective plate osteosynthesis procedure (clavicula, humerus, radius, ulna, femur, tibia, fibula, malleoli) (incl. delayed union, nonunion, malunion)
* Needed surgical instrument net: 2.4 / 2.7 / 3.5-4.0 / 4.5-5.0-6.5
* Adults (≥ 18 years)
* Written informed consent by patient

Exclusion Criteria:

* Bone disease (dysplasia's, sarcomas, chondroma's, osteolysis, osteomyelitis)
* Variable angle plates
* Corrective surgery after previous plate osteosynthesis procedure or hardware removal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Usability score of the ADEPTH sensor for bore depth measurements in plate osteosynthesis | Surgeon and OR assistant fill in the SUS after 3 operations in each study group. Anticipated study duration is 6 months.
  Used tool: System Usability Survey (SUS)

SECONDARY OUTCOMES:
Duration in seconds of the fixation process per screw during plate osteosynthesis | In both study groups the operation will be recorded. Anticipated study duration is 6 months.
  Tool: Video system in OR, video recording of each participant.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No